CLINICAL TRIAL: NCT03708523
Title: Next Day Early Morning Growth Hormone as Predictor of Pituitary Function After Transsphenoidal Adenomectomy
Brief Title: Next Day Growth Hormone Predicting Pituitary Function After Adenomectomy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201809035RIND
Record Dates: First submitted 2018-10-14; First posted 2018-10-17 (Actual); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Hypopituitarism
Keywords: Hypopituitarism,Pituitary function
MeSH Terms: conditions — Hypopituitarism

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study tried to highlight the predictive value of the morning postoperative cortisol levels, which can act as the prognosis value of the postoperative pituitary function, providing future medication advices for improving patients' safety of drugs.

DETAILED DESCRIPTION:
Transsphenoidal adenomectomy usually accompanied by the failure or recovery of the pituitary gland, which usually causing further hypopituitarism and hormone recovery. In order to prevent the potential applications of adrenal cortical malfunction after the surgery, many medical centers will use glucocorticoid supplements during the perioperative period care. However, this treatment might expose the normal hypothalamic-pituitary-adrenal (HPA) axis function patients into potential threats after the treatment of glucocorticoid supplements, such as bone loss, hypertension, emotional distress, and weight gain. To avoid unnecessary supply of glucocorticoids, the key question is to monitor the pituitary function. Thus, in this study we try to predict the morning postoperative cortisol levels, for further prediction of the postoperative pituitary function. To do so, we will review the retrospective charts of transsphenoidal adenomectomied patients from January, 2013 to April, 2018 in the NTUH Taipei. Use statistical methods analyzing all sorts of medical reports, including perioperative hormone thresholds.This study tried to highlight the predictive value of the morning postoperative cortisol levels, which can act as the prognosis value of the postoperative pituitary function, providing future medication advices for improving patients' safety of drugs.

ELIGIBILITY:
Inclusion:

Patients who had been treated with TSA were enrolled.

Exclusion:

1. Hypopituitarism preoperatively.
2. Acromegaly
3. Multiple operations
4. Incomplete hormone data or loss of follow-up

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who had been treated with TSA were enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2018-11-01 (Estimated); Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Next Day Early Morning Growth Hormone as Predictor of Pituitary Function After Transsphenoidal Adenomectomy | 2 days
  To predict the morning postoperative cortisol levels, for further prediction of the postoperative pituitary function.

CONTACTS AND LOCATIONS:
Overall Officials: Fon-Yih Tsuang, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan